CLINICAL TRIAL: NCT05469854
Title: A Phase I Study to Investigate the Pharmacokinetics and ECG Effects of Two Single Ascending Doses of Linaprazan Glurate Given as Oral Tablets to Healthy Subjects
Brief Title: A Study to Investigate the Pharmacokinetics and ECG Effects of Linaprazan Glurate
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cinclus Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CX842A2104
Record Dates: First submitted 2022-07-15; First posted 2022-07-22 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Pharmacokinetics; Cardiodynamic ECG; Safety, and Tolerability; GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linaprazan glurate (Experimental): Oral administration as a single dose of 300 mg, 600 mg, 200 mg, and a final dose level of maximum 400 mg.
  Interventions: Drug: Linaprazan glurate
- Placebo (Placebo Comparator): Oral administration as a singel dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linaprazan glurate — Linaprazan glurate base formulation, 25 mg oral tablets (300 mg and 600 mg doses).
  Linaprazan glurate hydrochloride (HCl), 25 mg and 100 mg (as base) oral tablets (200 mg and final dose level of maximum 400 mg).
  Other Names: X842
  Arms: Linaprazan glurate
Drug: Placebo — Single dose, oral tablets
  Arms: Placebo

SUMMARY:
This is a Phase I, single-center, double blind, placebo-controlled, parallel-group, randomized study designed to evaluate the PK, cardiodynamic ECG effects, safety, and tolerability of 2 single ascending oral doses of linaprazan glurate. The study will explore the PK properties of linaprazan glurate and linaprazan as well as the cardiodynamic ECG effects, safety, and tolerability after the administration of single doses (300 mg, 600 mg, 200 mg and a final dose level of maximum 400 mg) of linaprazan glurate, using 25 mg base formulation (300 mg and 600 mg doses) and 25 mg and 100 mg HCl formulation (200 mg and final dose level of maximum 400 mg) oral tablets.

ELIGIBILITY:
Main inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Healthy male or female aged 18 to 65 years
3. Body mass index ≥18.5 and ≤35.0 kg/m2.
4. Prospective subjects, as well as their partners, must agree to contraception requirements

Main exclusion criteria:

1. Female subjects of childbearing potential unless they agree to use highly effective methods of contraception (failure rate of <1%) from 2 weeks prior to dosing until the end-of-study visit.
2. Male subjects with a partner of childbearing potential, unless they agree to use method of contraception from 2 weeks prior to dosing until the end-of-study visit.History of or current clinically significant disease as defined in the protocol
3. History of or current clinically significant disease as defined in the protocol.
4. History of GERD, significant acid reflux.
5. Subjects who are pregnant, currently breastfeeding, or intend to become pregnant (female subjects) or father a child (male subjects) during the course of the study (i.e., from screening to end of study visit).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-12-02 (Estimated); Study Completion 2024-12-02 (Estimated)

PRIMARY OUTCOMES:
Measurement of pharmacokinetic profile of linprazan glurate and linaprazan (AUCinf) | Up to 24 hours
  To assess the Area under the plasma concentration vs. time curve (AUC) from time 0 to infinity (AUCinf)
Measurement of pharmacokinetic profile of linprazan glurate and linaprazan (AUClast) | Up to 24 hours
  To assess the AUC from time 0 to the last measurable concentration (AUClast)
Measurement of pharmacokinetic profile of linprazan glurate and linaprazan (Cmax) | Up to 24 hours
  To assess the Maximum plasma concentration (Cmax)
Measurement of pharmacokinetic profile of linprazan glurate and linaprazan (T1/2) | Up to 24 hours
  To assess the Terminal elimination half-life (T1/2)
Measurement of Cardiodynamic ECG (QTcF) | Up to 24 hours
  To assess the change from baseline in QTcF
Measurement of Cardiodynamic ECG (heart rate) | Up to 24 hours
  To assess the change from baseline in heart rate
Measurement of Cardiodynamic ECG (PR interval) | Up to 24 hours
  To assess the change from baseline in PR interval
Measurement of Cardiodynamic ECG (QRS interval) | Up to 24 hours
  To assess the change from baseline in QRS interval
Measurement of Cardiodynamic ECG (placebo-corrected QTcF) | Up to 24 hours
  To assess the change from baseline in placebo-corrected QTcF
Measurement of Cardiodynamic ECG (placebo-corrected heart rate) | Up to 24 hours
  To assess the change from baseline in placebo-corrected heart rate
Measurement of Cardiodynamic ECG (placebo-corrected PR interval) | Up to 24 hours
  To assess the change from baseline in placebo-corrected PR interval
Measurement of Cardiodynamic ECG (placebo-corrected QRS interval) | Up to 24 hours
  To assess the change from baseline in placebo-corrected QRS interval
Measurement of Cardiodynamic ECG (categorical outliers) | Up to 24 hours
  Number of categorical outliers for ECG parameters (QTcF, HR, PR interval, QRS interval)
Measurement of Cardiodynamic ECG (changes of T-wave) | Up to 24 hours
  Frequency of treatment emergent changes of T-wave abnormalities
Measurement of Cardiodynamic ECG (changes of U-wave) | Up to 24 hours
  Frequency of treatment emergent changes of U-wave abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rein-Hedin, MD, Principal Investigator — CTC Clinical Trial Consultants AB
Locations (1):
- CTC Clinical Trial Consultants AB, Uppsala, Sweden